CLINICAL TRIAL: NCT07099027
Title: The Lung Health Check Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LHC Pilot
Record Dates: First submitted 2025-05-06; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Screening; Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Health Check (Experimental): In this arm, consented participants will undergo a 'Lung Health Check' which incorporates a respiratory disease assessment, smoking cessation, low-dose CT and collection of biospecimens for translational analyses.
  Interventions: Diagnostic Test: Low dose CT

INTERVENTIONS:
Diagnostic Test: Low dose CT — In this arm, participants will undergo a respiratory assessment, smoking cessation, low-dose CT and biospecimen for translational research.

SUMMARY:
This study aims to test if it is feasible to introduce lung cancer screening in Ireland.

People within a certain age group, who smoke or who smoked in the past, are at a greater risk of developing lung cancer. They can also develop chronic lung conditions that can affect their long-term health. In Ireland, about 2,690 people are diagnosed with Lung Cancer every year. Unfortunately, 2 out of every 3 people diagnosed with lung cancer die per year.

The goal of this study is to try to screen for lung cancer in people before they have symptoms associated with the disease. We aim to do this by selecting people based on their age, whether they have smoked in the past or currently smoke as well as other relevant factors. People who take part in this study will have an assessment of how their lungs work and a low-dose CT scan. This is called a lung health check. The goal of the low-dose CT scan is to pick up lung cancer before it becomes symptomatic, and at an earlier stage. This scan uses a very low dose of radiation.

Unfortunately, without early detection, such as is the goal of this trial, 8 out of 10 people who go on to develop lung cancer will have advanced lung cancer when it is discovered, where outcomes tend to be poor. The earlier detection of lung cancer has a greater potential for treatment. Current international recommendations suggest carrying out these scans in the community rather than in a hospital. Therefore, we aim to deliver these lung health checks using a mobile unit in the community.

This study aims to test if we will successfully pick up lung cancer earlier by doing community-based 'lung health check's using mobile units in North Dublin and the North East, among people of a certain age and smoking history.

DETAILED DESCRIPTION:
Lung Cancer Screening Lung cancer is the leading cause of cancer-related death in both men and women, and leads to more deaths from cancer than breast, colon and prostate cancer combined(4). When a patient presents symptomatically with lung cancer, this is typically associated with advanced disease and poor survival. Using low-dose CT scan as a method of early detection to identify lung cancer in an at risk population, has been shown to reduce lung cancer mortality by 20-26% in two large clinical trials across the USA and Europe (5,6). The National Lung Cancer Screening Trial (NLST) was launched in 2002 across 33 centres in the USA. In total, almost 54,000 eligible participants were randomised to non-contrast enhanced computed tomography (CT) of the chest for three years versus postero-anterior chest x-ray (CXR). Eligible participants were selected based on clinical criteria, including: age 55-79; >30 pack-year smoking history; <15 years abstinence if former smoker, no history of other life-threatening cancers; no recent haemoptysis or weight loss indicative of lung cancer; no prior chest CT in the past year. The study demonstrated high compliance with screening low-dose CT with >90% of participants attending each annual visit. The study demonstrated a 20.3% relative reduction in lung cancer mortality (247 versus 309) per 100,000 person years with low-dose CT versus CXR. There was also a significant reduction in all-cause mortality by 6.7%. Significantly, low-dose CT was also associated with a 7% risk of an invasive follow-up procedure which resulted in a false positive (4% with CXR). A separate European study (The NELSON trial) investigated the use of low-dose chest CT annually for four years versus no screening in a randomised clinical trial reported in 2020 (5). In this study, eligible participants had to have smoked >15 cigarettes per day for >25 years or >10 cigarettes a day for >30 years. Participants were excluded if any of the following criteria were met: current or past renal cell cancer, melanoma, breast cancer; treatment related to lung cancer in the past 5 years; or a chest CT in the past year. This study did not exclude participants based on age alone. Due to accrual challenges amongst females, the primary endpoint analysis focused on 13,195 men which were randomised in this study. A further 2,594 women were included in the study and their outcomes were analysed as a secondary endpoint. This study demonstrated a significant reduction in lung cancer mortality in the screening group (156 vs. 206, HR = 0.76, 95% CI = 0.61 - 0.94). The incidence of false positives in this study was low (n=264/22,600, 1.2%). In summary, two large randomised controlled trials have demonstrated that low-dose CT scans of the chest reduce lung-cancer related mortality in high-risk participants.

A review of evidence by public health experts has revealed significant issues with attendance and implementation of early detection programs internationally. Targets in the United Kingdom for Breast and Bowel screening can be as low as 70% and 50% respectively. Evidence from UK studies show that barriers to uptake in screening programmes include a perceived lack of access to screening programmes and, a fatalistic attitude to lung cancer screening in deprived communities(7). In the UKLS trial, McDonald et al noted that the likelihood of lung cancer risk increased with socioeconomic deprivation but conversely response rates and clinic attendance fell (8). Reducing barriers to participation is a critical challenge to the implementation of early detection of lung cancer.

Spirometry and Lung Health Questionnaire While the large scale US (NLST) and European trials (NELSON) have provided sufficient evidence to show clinical efficacy, poor uptake and economic costs of lung cancer screening have led to significant difficulties with implementation to date. Particular issues include encouraging high-risk participants from socio-economically deprived areas to participate. However, researchers and clinical implementation groups in the UK have been leading initiatives aimed at addressing these logistical and deliverability issues through the launching of numerous implementation pilot trials that have led to the creation of high quality, pragmatic and cost-effective programmes. These studies have invited more than 500,000 participants, scanned 120,000 (24%) participants and diagnosed 15,000 lung cancers since 2019. Their widespread success has led to a recommendation by the UK National Screening Committee (UKNSC) to introduce a national lung cancer screening programme in the UK in 2023.

A cornerstone of the UK approach is the implementation of community-based screening, which has been to significantly improve attendance in pilot studies. Location and access to a dedicated CT scanner is fundamental to the success of these programmes. Access to CT scanning in hospital-based settings is at a premium and in order to facilitate high-volume scanning in participants to be assessed, access to a dedicated screening specific CT scanner is required. The seminal example of a successful UK based pilot 15 that has driven much of the further developments in national community based testing has been The Manchester Lung Health Check (LHC) pilot. This involved a community initiative which invited participants via their primary care team(9). The pilot programme invited participants aged 55-74 years, whom were ever smokers and were living in defined catchment areas of socioeconomic disadvantage. This study also used a validated lung cancer risk prediction model - PLCO2012(10). This prediction model incorporated clinical factors such as age, smoking history, pulmonary disease, family history etc. To be eligible for inclusion, participants needed to have a predicted risk of lung cancer >1.51%. Critically, the programme involved a community engagement initiative whereby the research study team engaged with persons in community centres and local organisations in order to educate and enhance awareness of the proposed screening pilot. The pilot study demonstrated an uptake of 28.5 % with a total 2827 participants attending the pilot. Of these 2827 participants, 49% (1384/2827) were eligible for low dose CT (LDCT) and proceeded to screening. A total of 3% (n=42) lung cancers were detected in this screening programme. This evidence indicates that a service that could identify people at high risk of lung cancer and provide them with a LDCT scan, would lead to a reduction in deaths from lung cancer. In the Manchester screening trial, they performed a comparative analysis of the PLCO2012 and LLPv2. In this study, they discovered that the LLPv2 was more sensitive at identifying participants with lung cancer in a deprived population(10). For this reason, we will use both scoring models in our proposed study.

Another successful UK based lung cancer screening pilot, the Yorkshire Lung Screening Trial (YLST) involved randomisation of eligible participants aged 55-80 to telephone based lung cancer risk assessment versus usual care(11) . In this study, a total of 44,393 participants were invited with an initial response rate of 50.8%. Amongst the respondents, 34.4% of participants were eligible and 86.8% of those underwent screening (n=6819). In this study, authors used a remote lung cancer risk assessment (telephone based). They demonstrated that telephone based risk assessment is a feasible strategy for a lung cancer screening pilot.

Lung Disease is one of the leading causes of premature mortality in Ireland. Approximately 20% of all respiratory deaths occur as a result of Chronic Obstructive Pulmonary Disease (COPD). Unfortunately, accurate data for the incidence and prevalence of COPD in the Irish participants is not available. However, approximately 50% of lifelong smokers will develop COPD at some stage in their lives (12). Estimates suggest about 500,000 participants in Ireland may have COPD of whom 200,000 potentially have moderate and severe forms of disease. It is estimated that between 30-50% of these participants are currently undiagnosed. Late or underdiagnosed COPD is a significant health and health economic burden to the state with a strong association with hospital admissions for exacerbations. Approximately 30% of participants who present to hospital emergency departments with emergent COPD have had no formal diagnosis(13). Ireland also has the highest rate of hospital admission for COPD exacerbation in the OECD and the Beaumont Hospital catchment area has one of the highest rates of hospital admission for COPD exacerbation in the country at 376 admissions per 100,000 participants. The rate of decline in lung function is also faster in the earlier stages of the disease and therefore the potential for altering the course of the disease and improving outcomes is greater when identified earlier and when correct treatment interventions are initiated. Selected published lung cancer screening studies, where spirometry is performed, have shown that approximately 10-15% of lung cancer screening attendees have undiagnosed symptomatic COPD. As yet the data is unclear if routine spirometry improves health outcomes for lung cancer screening participants, but it is an area that warrants significant investigation and a Lung Health Check (LHC) environment is well-placed to enable such investigations. Spirometry may also help further stratify lung cancer risk in these participants as it acts as evidence of airway obstruction, which is an independent risk factor for the development of lung cancer.

Smoking Cessation Smoking cessation is an essential component of any lung cancer screening pilot trial or programme. The UKLS trial showed that lung cancer screening, particularly when associated with an abnormal scan result increases smoking cessation rates and represents a powerful opportunity to maximise smoking cessation rates. Cost-effectiveness data also shows that adding smoking cessation interventions is cost-effective, resulting in additional cancer deaths averted and life-years gained compared with screening alone. UK-based models of delivery advise that smoking cessation should be delivered by an opt-out approach, to reduce stigmatisation and should involve a co-located smoking cessation practitioner who is able to provide a comprehensive package of smoking cessation supports in an immediate fashion. UK policy advice suggests that consideration should be given to the use of Nicotine replacement therapy (NRT) as well as electronic cigarettes and vaping devices.

In summary, the evidence indicates that a service to identify people at high-risk of lung cancer and provide them with a low-dose chest CT scan would lead to a reduction in deaths from lung cancer. Equally, lung cancer screening is only effective with sufficient 16 uptake amongst high-risk participants. Experience internationally (e.g. Manchester LHC) would suggest the need for pilot studies to ensure adequate community engagement in lung cancer screening. We thus propose the first pilot study of lung cancer screening in Ireland, using a GP-referral mechanism, remote PLCO scoring, and attendance at a community-based LHC facility incorporating spirometry, smoking cessation and a low-dose CT scan of the chest.

The "Lung Health Check Pilot (LHC Pilot)" aims to provide a free low-dose CT scan to high-risk participants in an area with a high burden of lung cancer (North Dublin/North East Region). A pilot early detection program will be designed to minimise barriers to participation by:

1. maximizing convenience through use of a community-based LHC/CT scan unit
2. placing it strategically in a high prevalence area (North Dublin/North East Region) with high footfall or easy accessibility
3. Incorporating supportive measures to maximise favourable outcomes in this participants through a respiratory assessment, and the incorporation of smoking cessation, as part of the LHC pilot.

We will also embed a translational research aims in this pilot study, to create a biorepository of breath and blood samples from participants to inform the next generation of lung cancer early detection methods and future prevention clinical trials through identification of non-invasive biomarkers.

High-risk participants (ever-smokers, aged 55-74 years) will be identified via GP practice databases and invited to undergo a 'lung health check'. As GP data is likely to be incomplete in this regard, invitations will be extended to all adults aged 55-74 years using low burden patient information leaflets and a dedicated invitation via an approved third-party vendor. These leaflets will be initially sent to each patient informing them of the pilot study, its benefits and who it is designed for. A formal letter of invitation will then be sent shortly after. Participants will be invited to participate via phonecall and letter. Participants who are invited to take part will be contacted via phoneline by qualified personnel, and asked an initial set of questions ensuring the participant is eligible to participate in the study based on the outlined inclusion and exclusion criteria (see section 2.6), and completion of their Validated PLCO (m2012) score (calculated cut-off point of 1.51%) and LLPv2 score (cut-off ≥2.5%). If they are eligible based on these assessments by phone, they will be invited to attend an in-person LHC at the community-based site, that includes a low dose CT chest(10) at a designated time. Those with a negative lung cancer risk assessment will be deemed not eligible to participate, and will be discharged from the programme via return letter. For those who attend the LHC, screening visits will be offered over two rounds, one year apart. Any identified pulmonary nodules on LHC performed CT will be analysed according to BTS pulmonary nodule guidelines and categorized as negative, indeterminate or positive. A case of suspected lung cancer (positive results) will require immediate referral to the local rapid access lung clinic, while indeterminate results will have an initial 3-month surveillance CT scan. CT reporting will be carried out by a group of radiologists with interest, expertise and training in Thoracic Oncology and BTS guidelines. Clinically-relevant incidental findings that require further clarification or work-up will be referred for GP or hospital specialist review and/or be discussed at a monthly dedicated Screening MDT in the Beaumont Hospital before deciding management plan. Some pulmonary nodules that need further discussion before follow-up planning will be discussed at this meeting also. The meeting will be attended by at a minimum: a respiratory Physician, a thoracic radiologist and the LHC programme manager.

The study will aim to 1) Explore the feasibility of a Lung Health Check (LHC) programme which incorporates a LDCT, respiratory disease assessment, and smoking cessation advice, in Ireland; 2) Identify the incidence, stage, treatment and outcomes of participants diagnosed with lung cancer in the high-risk participants; 3) Assess tobacco dependency of the high-risk participants with, reassessment after a community-based smoking cessation programme; 4) Define the proportion of participants with known or newly diagnosed respiratory disease and their management, as part of the LHC pilot; 5) Identify breath and blood-based biomarkers in participants; 6) Identify the optimal mechanism for the assessment eligibility for lung cancer screening in Ireland.

ELIGIBILITY:
Inclusion Criteria:

1. 55 - 74 years of age
2. Current or former smokers

   * Current: >100 cigarettes in lifetime and/or currently tobacco smoking
   * Former: >100 cigarettes in lifetime and/or no tobacco smoking >= 28 days
3. Referred from a GP for the LHC pilot
4. PLCOM2012 ≥ 1.51% or LLPv2 ≥2.5% (Lung Cancer Risk Scores)

   * Prostate Lung Cancer Colorectal Ovarian (PLCO) & Liverpool Lung Project Version 2 (LLPv2)

Exclusion Criteria:

1. Participant-reported history of chest CT in the last 12 months
2. Inability to undergo non-contrast CT (e.g. >200 kg body weight, inability to lie flat)
3. Participant reported known diagnosis of other advanced stage cancers
4. Participant reported diagnosis of lung cancer of any stage in the last 5 years
5. Likely non-compliance with study procedures, as determined by the participant i) Unable to provide informed consent ii) Inability to attend study visits
6. Nursing home residents -

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2183 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
i) The proportion of high-risk eligible participants aged 55-74 years who participate in a community-based lung health check ii)The proportion of individuals who consent to undergo telephone assessment | 1 year
  i) Number of eligible participants who attend the LHC pilot after GP invitation/Number of high-risk participants invited via GP letter to the LHC pilot ii) Number of participants who consent to undergo telephone assessment/number of participants invite via GP letter to LHC pilot
The proportion of individuals who consent to undergo telephone assessment | 1 year
  Number of individuals who consent to undergo telephone assessment/Number of individuals invited via GP letter to the LHC pilot ii) Number of participants who consent to undergo telephone assessment/number of participants invite via GP letter to LHC pilot

SECONDARY OUTCOMES:
The proportion of the participants (aged 55-74 years, from catchment area, who receive GP invitation) who attend a community-based initial (T0)LHC visit, and the mandated follow-up visit (T1) | 2 years
  The proportion of the participants (aged 55-74 years, from catchment area, who receive GP invitation) who attend a community-based initial (T0)LHC visit, and the mandated follow-up visit (T1)
The proportion of participants (aged 55-74 years, from catchment area, who receive GP invitation) who attend a community-based T0 LHC visit, that are deemed eligible to participate based on eligibility criteria and risk scores | 1 year
  The proportion of participants (aged 55-74 years, from catchment area, who receive GP invitation) who attend a community-based T0 LHC visit, that are deemed eligible to participate based on eligibility criteria and risk scores
The proportion of high-risk eligible participants aged 55-74 years for whom an appointment is booked in a community-based LHC visit | 1 year
  The proportion of high-risk eligible participants aged 55-74 years for whom an appointment is booked in a community-based LHC visit
The proportion of high-risk participants that attend from an urban versus rural setting. | 1 year
  The proportion of high-risk participants that attend from an urban versus rural setting.
The proportion of high-risk participants that respond to the LHC invitation and are deemed eligible by age, gender, socioeconomic status, social deprivation index, and presence of co-morbid conditions | 1 year
  The proportion of high-risk participants that respond to the LHC invitation and are deemed eligible by age, gender, socioeconomic status, social deprivation index, and presence of co-morbid conditions
The proportion of high-risk participants that attend the LHC, by age, gender, socioeconomic status, social deprivation index, and presence of co-morbid conditions | 1 year
  The proportion of high-risk participants that attend the LHC, by age, gender, socioeconomic status, social deprivation index, and presence of co-morbid conditions
The proportion of participants who attend the initial screening round who attend subsequent screening rounds (T0+3/T1) | 1 year
  The proportion of participants who attend the initial screening round who attend subsequent screening rounds (T0+3/T1)
Number of participants referred to the Hospital Rapid Access Lung Cancer Clinic (RALCC) as a result of the LHC. | 3 years
  Number of participants referred to the Hospital Rapid Access Lung Cancer Clinic (RALCC) as a result of the LHC.
Number of participants referred to the Beaumont Hospital Lung Cancer MDT as a result of the LHC. | 3 years
  Number of participants referred to the Beaumont Hospital Lung Cancer MDT as a result of the LHC.
Proportion of participants that attend a LHC visit who are subsequently diagnosed with lung cancer. | 3 years
  Proportion of participants that attend a LHC visit who are subsequently diagnosed with lung cancer.
Proportion of participants with lung cancer who are diagnosed with earlier stage lung cancer (stage I/II vs stage III/ IV), compared with national registry data on initial stage at diagnosis in the last 5 years. | 4 years
  Proportion of participants with lung cancer who are diagnosed with earlier stage lung cancer (stage I/II vs stage III/ IV), compared with national registry data on initial stage at diagnosis in the last 5 years.
Proportion of participants diagnosed with lung cancer, who receive lung cancer treatment by modality and treatment intention (e.g. surgery, radiation therapy, systemic therapy; curative vs. palliative) | 3 years
  Proportion of participants diagnosed with lung cancer, who receive lung cancer treatment by modality and treatment intention (e.g. surgery, radiation therapy, systemic therapy; curative vs. palliative)
The proportion of high-risk participants diagnosed with lung cancer who have a: i) PLCOm2012 ≥ 1.51% ii) LLPv2≥2.5%* | 3 years
  The proportion of high-risk participants diagnosed with lung cancer who have a:
  i) PLCOm2012 ≥ 1.51% ii) LLPv2 ≥2.5%*
Number of participants with incidental findings identified on low-dose CT | 4 years
  Number of participants with incidental findings identified on low-dose CT
Number of participants with newly diagnosed COPD from baseline spirometry and respiratory health questionnaires, complete as part of the LHC | 4 years
  Number of participants with newly diagnosed COPD from baseline spirometry and respiratory health questionnaires, complete as part of the LHC
Nodule Detection Rate: The percentage of participants who have one or more nodules detected during the LHC (Nodule definition as per BTS Guidelines(1) | 4 years
  Nodule Detection Rate: The percentage of participants who have one or more nodules detected during the LHC (Nodule definition as per BTS Guidelines(1)
Nodule Size: Nodule size for all nodules reported on T0 LHC CT | 4 years
  Nodule Size: Nodule size for all nodules reported on T0 LHC CT
Nodule Growth Rate: For all patients with >1 CT scan and >=1 nodule. Growth rate will be defined and recorded. (Nodule Size at Follow-up CT/Nodule Size from CT at T0). | 4 years
  Nodule Growth Rate: For all patients with >1 CT scan and >=1 nodule. Growth rate will be defined and recorded. (Nodule Size at Follow-up CT/Nodule Size from CT at T0).
False-Positive Rate: The percentage of participants who are investigated through RALCC for a suspicious nodule/suspected lung cancer that turns out to be non-malignant after investigation. | 4 years
  False-Positive Rate: The percentage of participants who are investigated through RALCC for a suspicious nodule/suspected lung cancer that turns out to be non-malignant after investigation.
False-Negative Rate: The percentage of participants who are investigated through RALCC for a suspicious nodule/suspected lung cancer that turns out to be non-malignant after investigation. | 4 years
  False-Negative Rate: The percentage of participants who are investigated through RALCC for a suspicious nodule/suspected lung cancer that turns out to be non-malignant after investigation.
Interval Cancer: a lung cancer diagnosed following a symptomatic presentation between screening rounds "outside screening," | 4 years
  Interval Cancer: a lung cancer diagnosed following a symptomatic presentation between screening rounds "outside screening,"
Sensitivity (True positive cases) | 4 years
  Sensitivity (True positive cases)
Specificity (True-negative cases) | 4 years
  Specificity (True-negative cases)
Referral rate: The percentage of participants referred for further investigation due to an incidental finding that requires medical assessment by either the participant's GP or a hospital specialist | 4 years
  Referral rate: The percentage of participants referred for further investigation due to an incidental finding that requires medical assessment by either the participant's GP or a hospital specialist
Identify participant smoking rates before and after a brief smoking intervention followed by opt-out referral to HSE led community-based smoking cessation programme for current smokers, as part of the LHC. | 4 years
  Identify participant smoking rates before and after a brief smoking intervention followed by opt-out referral to HSE led community-based smoking cessation programme for current smokers, as part of the LHC.
Proportion of participants who participate in the HSE led opt-out smoking cessation programme, after participation in the LHC pilot. | 4 years
  Proportion of participants who participate in the HSE led opt-out smoking cessation programme, after participation in the LHC pilot.
1-year smoking cessation rates at T1 vs. T0 timepoints. | 4 years
  1-year smoking cessation rates at T1 vs. T0 timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Jarushka Naidoo, MD, Principal Investigator — Beaumont RCSI Cancer Centre
Locations (1):
- Beaumont RCSI Cancer Centre, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O Reilly D, Roche S, Noonan C, O'Shea J, Toomey S, Hennessy BT, Fitzmaurice GJ, Egan K, Dunne J, Dowling CM, Counihan I, O'Brien E, Sulaiman I, Morgan R, Jacob B, Baird AM, Cotter S, Bailey D, Maguire G, Bennett K, Sorensen J, Healy NA, Ryan J, Redmond P, Ryan DJ, Naidoo J. Lung Health Check pilot: Ireland's flagship lung cancer screening trial. BMJ Open Respir Res. 2025 Sep 10;12(1):e003035. doi: 10.1136/bmjresp-2024-003035. PMID 40935563
- See also: Lung Heath Check website — https://lunghealthcheck.ie/